CLINICAL TRIAL: NCT01883258
Title: Mechanisms of Cardiovascular Dysfunction and Effect of Aerobic Exercise Training in Adults With Type 2 Diabetes
Brief Title: Effect of Aerobic Interval Training on Cardiovascular Function in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB201601534-N; 280-2012 (Other: Legacy study); 1R21AG050203-01 (NIH); OCR12584 (Other: University of Florida)
Record Dates: First submitted 2013-06-13; First posted 2013-06-21 (Estimated); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High intensity aerobic interval training (Experimental): Type 2 diabetes subjects will complete 8 weeks of high intensity aerobic interval exercise training.
  Interventions: Other: High intensity aerobic interval training
- Continuous moderate intensity exercise (Experimental): Type 2 diabetes subjects will complete 8 weeks of continuous moderate intensity exercise training.
  Interventions: Other: Continuous moderate intensity exercise
- Non-exercise control group (No Intervention): Type 2 diabetes subjects assigned to the non-exercise control group will maintain their normal lifestyle for 8 weeks.
- Healthy control group (No Intervention): Healthy subjects will be assigned to the healthy control group and will undergo baseline measures only.

INTERVENTIONS:
Other: High intensity aerobic interval training — Supervised aerobic interval training will be performed on bicycles 4 times per week for 8 weeks. Each training session will last 40 minutes and will consist of 10-minute warm up at 70% of maximal heart rate (HRmax), four 4-minute intervals at 90% of HRmax with 3-min active recovery at 70% of HRmax and 5-minute cool down at 70% of HRmax.
  Arms: High intensity aerobic interval training
Other: Continuous moderate intensity exercise — Supervised exercise training will be performed on bicycles 4 times per week for 8 weeks. Each training session will last 47 minutes and will consist of continuous moderate intensity cycling at 70% of HRmax.
  Arms: Continuous moderate intensity exercise

SUMMARY:
The study objectives are:

1. To compare cardiovascular function in type 2 diabetes patients vs. healthy controls.
2. To compare the effect of 8 weeks of aerobic interval training versus continuous moderate exercise on cardiovascular function in adults with type 2 diabetes.
3. To examine the mechanisms underlying the exercise-related changes in cardiovascular function.

The investigators hypothesize that compared to continuous moderate intensity exercise training, interval training will be more effective in improving cardiovascular function in adults with type 2 diabetes.

DETAILED DESCRIPTION:
Cardiovascular function will be measured at baseline in adults with type 2 diabetes and in age-matched healthy controls. Research volunteers with type 2 diabetes who meet the inclusion criteria will be randomized to the aerobic interval training group, continuous moderate exercise group or non-exercise control group. At the end of the 8-week randomized control exercise intervention, baseline measures will be repeated.

ELIGIBILITY:
Inclusion Criteria for type 2 diabetes :

* Diagnosis of type 2 diabetes
* Sedentary or minimally physically active for at least the prior 1 year
* Able to give consent

Inclusion criteria for healthy control group:

* Sedentary or minimally physically active for at least the prior 1 year
* Able to give consent

Exclusion Criteria:

* History of diabetic proliferative retinopathy, autonomic or peripheral neuropathy
* History of any relevant cardiovascular diseases (myocardial infarction, angina pectoris, history of coronary artery bypass surgery or angioplasty, congestive heart failure, or arrhythmia)
* Hypertension (≥160 mmHg systolic or ≥100 mmHg diastolic)
* History of renal impairment
* History of gout or hyperuricemia
* History of hepatic disease or infection with hepatitis B, C
* History of seizures, or other relevant on-going or recurrent illness
* Recent (within 3 months) or recurrent hospitalizations
* Use of tobacco products
* >5 % weight change in the prior 6 months.
* Current intake of medications that may affect study results
* Premenopausal women taking oral contraceptives and postmenopausal women taking hormone replacement therapy.
* Pregnancy (positive urine pregnancy test) or lactation
* For the healthy control group, history of diabetes.

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2018-07-16 (Actual); Study Completion 2018-07-16 (Actual)

PRIMARY OUTCOMES:
Change in vascular endothelial function | At baseline and after 8 weeks of exercise training
  Brachial flow mediated dilation using ultrasonography

SECONDARY OUTCOMES:
Change in factors related with endothelial function | At baseline and after 8 weeks of exercise training
  Blood and cellular markers of adiponectin, oxidative stress and inflammation.
Change in arterial stiffness | At baseline and after 8 weeks of exercise training
  Arterial stiffness (pulse wave velocity) and wave reflection (augmentation index) will be measured using the SphygmoCor device.
Change in cardiac function | At baseline and after 8 weeks of exercise training
  Left ventricular systolic and diastolic function will be measured using echocardiography.
Change in maximal oxygen consumption | At baseline and after 8 weeks of exercise training
  Maximal oxygen consumption will be measured using online computer-assisted open-circuit spirometry during incremental treadmill exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Demetra D Christou, Ph.D, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States